CLINICAL TRIAL: NCT02851537
Title: Magnetic Resonance Spectroscopy at Term-equivalent Age and Executive Functions at 5 Years of Age Corrected in Very Preterm Infants
Acronym: EPIRMEX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-17
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Children Born Very Prematurely in Relation to Structural Brain Abnormalities
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: an advanced technique as magnetic resonance spectroscopy (MRS) — subjects who had an advanced technique as magnetic resonance spectroscopy (MRS) It is based on the detection of cerebral metabolites, and the variations of their concentration to characterize different pathologies.

SUMMARY:
EPIRMEX is a complementary study to the national cohort EPIPAGE 2 the INSERM Unit 953 is responsible. The objective of this study is to evaluate at the age of 5 years corrected executive functions in children born very prematurely in relation to structural brain abnormalities in magnetic resonance imaging (MRI) (technical conventional and advanced) performed at the age of term. The current study is a project on a subset of the population of premature EPIRMEX subjects who had an advanced technique as magnetic resonance spectroscopy (MRS). It is a recent imaging technique for a study of the cerebral metabolism. It is based on the detection of cerebral metabolites, and the variations of their concentration to characterize different pathologies. In most cases, combinations of metabolites are informed creatine + phosphocreatine (CR), glycerophosphocholine + phosphocholine (CHO) + Nacétylaspartate Nacetylaspartylglutamate (NAA), myoinositol (INS) and lactate (LAC). In the premature newborn, the NAA / CHO ratio increases with age in all brain regions. The LAC / NAA ratio decreases significantly with age in the thalamus, basal ganglia, the corticospinal tract, and parietal white matter tends to decrease elsewhere . A number of studies show that proton spectroscopy term can predict the long-term newborn who presented an anoxic-ischemic encephalopathy .These studies indicate that an increase in lactate and a decrease in NAA are correlated with abnormal neurological development. And decreases in NAA / CR and / or NAA / CHO ratios are predictive of motor abnormalities in children with anoxic encephalopathy presented an ischemia . These decreases were also measured in the basal ganglia, occipital cortex, and areas near the last. Few studies have explored the magnetic resonance spectroscopy of proton-term prediction of the future of large premature.

DETAILED DESCRIPTION:
This is a prospective cohort study on a subsample of children born prematurely (before 33 weeks of gestation (SA) otherwise included in the national cohort EPIPAGE 2 and included in epirmex and who enjoys a spectrosocpie. This research project proposed in the framework of the AORC as ancillary study EPIPAGE 2 -EPIRMEX therefore focuses on spectroIRM voluntarily at the age of term (39-41 SA), and more specifically the emergence executive functions to 5 years EPIRMEX main objective of the study. the application of our project to this tender is requested by the PACA region due to the high rate spectroIRM performed by our area (about 75%) and strong involvement of Dr. C. Gire in EPIPAGE 2 and EPIRMEX. However, only neuropsychological assessments FE 5 years testing sub-cities will be funded EPIPAGE 2. The specific aspect of our study is not funded EPIPAGE 2.

The children received conventional MRI at the age of term (39-41 SA), supplemented by specific sequences for single voxel analysis in microstructural analysis (white matter, basal ganglia and brainstem), short echo and echo time consuming. The study of the spectra will be done quantitatively by CEMEREM laboratory - UMR 6612 CNRS / Université de la Méditerranée / Division of Medical Imaging (Pr Guye).

The relevance of the project was its ability to include quality as 550 MRI were performed, including 120 MRI spectrometer can be analyzed.

These children were assessed within 2 EPIPAGE the corrected age of 2 years, 3 years (EPIRMEX) and 5 years (2 + EPIPAGE EPIRMEX). The balance sheet under 5 years in EPIRMEX is evaluating a comprehensive intellectual efficiency WPPSI III, some elements of the NEPSY and the figure of REY.

So magnetic resonance spectroscopy may provide additional diagnostic value to cranial ultrasound and MRI in infants.

The main objective is to assess the relation between the cerebral MRS at term-equivalent age of very preterm infants and the executive functions at the age of 5 years corrected.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 26+ 0d and 32 SA + 6d.
* Children included in the study EPIPAGE2, and EPIRMEX and has received spectroscopy.
* Regions of interest analyzed: periventricular area, basal ganglia, brain stem.
* Who has full cognitive assessment in epirmex to 5 years.

Exclusion Criteria:

* Children with severe chromosomal anomaly.
* Children with central nervous system malformation diagnosed prenatally or on examinations in the neonatal period (transfontanellaire ultrasound and/or MRI).

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children born very prematurely in relation to structural brain abnormalities and has received spectroscopy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
assessment of the executive dysfunction | one day
  NEPSY score <-1 DS is <8 (required) it is a tool to assess the neuropsychological development of children of preschool and school age (3 to 12 years)
intellectual efficiency | one day
  Wechsler Preschool and Primary Scale of Intelligence (WPPSI)
perceptual organization and memory | one day
  figure of REY is a short test of perceptual organization and memory. The figure of Rey is called abnormal for a copy <10th percentile.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille